CLINICAL TRIAL: NCT03990103
Title: S1 Plus Paclitaxel (IV&IP) Plus Bevacizumab (IP) Versus S1 Plus Oxaliplatin(IV) as First-line Treatment in Gastric or Gastroesophageal Junctional Adenocarcinoma With Malignant Ascites: An Open-label, Multicenter Phase II Study
Brief Title: S1+ Paclitaxel (IV&IP) + Bevacizumab (IP) Versus S1+Oxaliplatin as First-line Treatment in Gastric Cancer With Malignant Ascites
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director, China Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOG1704
Record Dates: First submitted 2019-05-28; First posted 2019-06-18 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Gastric Adenocarcinoma
Keywords: Gastric Carcinoma; Malignant Ascites; Intraperitoneal Chemotherapy; Bevacizumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Paclitaxel; Bevacizumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): S1+Paclitaxel (IV&IP)+Bevacizumab (IP)
  Interventions: Drug: S1; Drug: Paclitaxel; Drug: Bevacizumab
- Control arm (Active Comparator): S1+Oxaliplatin (IV)
  Interventions: Drug: S1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: S1 — 80-120 mg/day, PO, D1-14, every 21 days
  Other Names: Tegafur Gimeracil Oteracil Potassium Capsule
Drug: Paclitaxel — 20 mg/m2/day, IP, D1-3; 50 mg/m2, IV, D1; 70 mg/m2, IV, D8; every 21 days
  Other Names: Paclitaxel Injection
  Arms: Experimental arm
Drug: Bevacizumab — 200 mg, IP, D1, every 21 days
  Other Names: Avastin ®
  Arms: Experimental arm
Drug: Oxaliplatin — 130 mg/m2, IV, D1, every 21 days
  Other Names: ELOXATIN®
  Arms: Control arm

SUMMARY:
The purpose of this study is to compare the efficacy of S1 plus paclitaxel (intravenous injection & intraperitoneal injection) plus bevacizumab (intraperitoneal injection) vs. S1 plus oxaliplatin intravenous injection as first-line treatment in gastric or gastroesophageal junctional adenocarcinoma with malignant ascites.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter clinical trial, to compare the efficacy of S1 plus paclitaxel (intravenous injection & intraperitoneal injection) plus bevacizumab (intraperitoneal injection) versus S1 plus oxaliplatin intravenous injection as first-line treatment in gastric or gastroesophageal junctional adenocarcinoma with malignant ascites. A total of 66 patients who are diagnosed with gastric or gastroesophageal junctional adenocarcinoma will be allocated to receive either S1 orally administration plus paclitaxel intravenous injection & intraperitoneal injection plus bevacizumab intraperitoneal injection, or to receive S1 orally administration plus oxaliplatin intravenous injection. The primary end point is ascites response rate at 6 weeks. The secondary end points include the median overall survival (OS), progression-free survival (PFS), time to treatment failure (TTF), objective response rate (ORR), puncture free survival, volume of drainage, the quality of life (QoL) and safety.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≥ Age≤ 70 years, male or female
* Pathologically confirmed adenocarcinoma of the gastric or gastro-oesophageal junction with inoperable locally advanced or recurrent and/or metastatic disease; with medium amount of malignant ascites which can be catheterized.
* Diagnostic criteria for malignant ascites (meet any of the following criteria): ascites cytology positive; or imaging or pathological confirmed peritoneal metastases.
* No prior anti-tumor treatment to the metastatic disease; an interval of at least 6 months from the last adjuvant chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status( PS) score 0-1.
* Normal major organ function, and laboratory tests must meet the following criteria: hemoglobin (HGB) ≥ 90 g/L, neutrophil count ≥ 1.5×109/L, platelet count ≥ 100×109/L, total bilirubin (TBil) ≤ 1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 UNL, serum creatinine (Cr) ≤ 1 UNL; creatinine clearance rate (CCr) ≥ 60 ml/min (calculated using the Cockcroft-Gault equation).
* International Normalized Ratio (INR) ≤ 1.5 and partial prothrombin time (PPT) or activated partial thromboplastin time (APTT) ≤ 1.5 UNL within 7 days before enrollment.
* Life expectancy of at least 12 weeks
* Signed informed consent (ICF)
* For women of child bearing potential, a negative serum or urine pregnancy test result should be obtained with 7 days before enrollment; Women of childbearing potential and men must agree to use adequate contraception before entering the program until at least 8 weeks after the last study drug administration.

Exclusion Criteria:

* Known hypersensitivity or allergic to any of the study drugs, study drug classes, or excipients in the formulation.
* Subject received chemotherapy to the metastatic disease (except adjuvant/neoadjuvant chemotherapy administered 24 weeks before enrollment)
* Subject with other malignancies, except for non-melanoma skin cancer or in-situ cervical carcinoma under adequate treatment, or other treated malignancies without evidence of recurrent for 5 years.
* Anti-tumor cytotoxic drug therapy within 14 days prior to enrollment（longer washout time interval might needed depends on drug characteristics）
* Uncontrolled hypertension which cannot be reduced to normal range by antihypertensive agents [Systolic Blood Pressure(SBP) >140 mmHg, diastolic blood pressure (DBP) > 90 mmHg], coronary artery disease > grade 1, arrhythmia > grade 1 [including corrected QT(QTc) interval prolongation: QTc>450 ms for male，QTc>470 ms for female], grade 1 heart failure.
* Proteinuria ≥ ++，or persistent proteinuria > 1.0 g/24 hours
* Presence of any toxicity ≥ grade 1 according to NCI-CTCAE except for alopecia.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks, cerebral hemorrhage、cerebral infarction), deep vein thrombosis and pulmonary embolism within 12 months before enrollment.
* Bowel obstruction within 6 weeks before enrollment.
* Surgical treatment was performed within 6 weeks before enrollment. Subject should recover from any major surgery.
* Serious uncontrolled systemic illness or medical condition or uncontrolled infections, including but not limited to: uncontrollable ventricular arrhythmias, history of documented myocardial infarction within 3 months, uncontrollable epileptic dementia, unstable spinal compression, superior vena cava syndrome, extensive bilateral interstitial pulmonary disease by high-resolution computed tomography (HRCT), or any neurological or mental abnormalities which affect compliance.
* Human immunodeficiency virus (HIV) positive
* Pregnancy or lactation women
* Cannot be orally administered medication
* Subject with a tendency for gastrointestinal hemorrhage. Including: Black stool or hematemesis within 2 months; For subjects positive in occult test with unresected primary lesion, if the principle investigator in each center considers with possibility of gastrointestinal hemorrhage, the subject could not be enrolled.
* Subject with malignant pleural effusion need medical intervention.
* A history or evidence of hereditary hemorrhagic constitution or coagulation disorder that increases the risk of bleeding
* Subjects with central nerve system metastases
* Have been enrolled in other clinical trial with investigational drug treatment within the 4 weeks of start of study treatment
* For subject with bone metastases, palliative radiotherapy was given 4 weeks before enrollment (radiation field >5%).
* Any other disease or condition that the investigator considers not suitable for participating in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Ascites response rate at 6 weeks | 6 weeks
  response of ascites at 6 weeks

SECONDARY OUTCOMES:
PFS | 12 months
  Progression-free survival,From 1st drug administration to the date of first progression or date of death (whichever occurs first)
OS | 2 years
  Overall survival, from enrollment until death from any cause
ORR | 12 months
  Objective response rate, the proportion of patients with reduction in tumor burden of a predefined amount
TTF | 12 months
  Time to treatment failure, from 1st drug administration to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death
Puncture free survival | 12 months
  Puncture free survival time, from the first puncture to secondary puncture
Volume of drainage | 12 months
  Volume of drainage
Adverse events | 12 months
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, M.D., Principal Investigator — China Medical University, China
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided